CLINICAL TRIAL: NCT01197118
Title: Phase 2 Study of Chemoradiotherapy for Advanced Gastric Cancer
Brief Title: Postoperative Sequence Chemoradiotherapy Compared With Chemotherapy Alone for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Shiying Yu / Chief, Tongji Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJCC-GC001
Record Dates: First submitted 2009-04-23; First posted 2010-09-09 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; sequence chemoradiotherapy; OLF regimen; survival rate
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): chemotherapy alone following radical resection
  Interventions: Drug: chemotherapy alone following radical resection
- 1 (Experimental): sequence chemoradiotherapy following radical resection
  Interventions: Radiation: sequence chemoradiotherapy

INTERVENTIONS:
Radiation: sequence chemoradiotherapy — Postoperative radiotherapy regimen: Therapy plan system was formulated by Computed tomographic (CT) simulation. Radiation was delivered with 15MV photons. Radiotherapy consisted of 4500 cGy of radiation at 180 cGy per day, five days per week for five weeks, to the tumor bed, to the margins of resection or the stoma, to the regional nodes. Protection of spinal cord, heart, liver and kidney should be considered.
  Postoperative chemotherapy regimen: see arm 2
  Arms: 1
Drug: chemotherapy alone following radical resection — Postoperative chemotherapy regimen: The OLF regimen was administrated: Oxaliplatin, 130 mg/m2/day on day1, i.v. 2 h; fluorouracil, 425 mg/m2/day on day1~5, i.v.; leucovorin, 200 mg/m2/day on day 1~5, i.v.; every 21 days repeated, for 6 cycles.
  Arms: 2

SUMMARY:
Gastric cancer is one of the most prevalent malignancies in China; the survival rate remains poor despite potentially curative resections. Complete surgical resection is the only potentially curative therapy available to patients with gastric cancer. However, even after a complete resection with negative margins, many patients will experience recurrence. In recent years, the radiation therapy in the carcinoma of the stomach represents a new issue that should be addressed accompanying the development of radial physics and radial biology, the clinical application of computed tomographic (CT) simulation and digital reconstitution technique, especially the application of 3-dimensional conformal and intensity modulated radiation therapy. Radiation therapy plus concurrent chemotherapy has been demonstrated to cause a significant improvement in overall and disease-free survival according to Intergroup Trial 0116/SWOG 9008. So the investigators designed the trial to see whether a postoperative sequence chemoradiotherapy including oxaliplatin fluorouracil-based regimen can improve survival for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Postoperative histologically confirmed advanced adenocarcinoma of the stomach or the gastroesophageal junction.
2. Age of 18 to 75, Karnofsky score higher than 70.
3. Postoperative histologically conformed metastasis in perigastric lymph nodes and/or tumor invasion to muscularis propria or subserosa, with or without positive incisal margin.
4. No severe functional damage of major organ, normal blood cell, normal liver and kidney function.
5. No clinical findings of distant metastasis.
6. Predictive survival time longer than 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shiying Yu, Master, Principal Investigator — Tongji Cancer Center
Locations (1):
- Tongji Cancer Center,Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Xiang-Lin Yuan, Qiang Fu ,Shi-Ying Yu .Postoperative sequence chemoradiotherapy for advanced gastric cancer:an analysis of 36 cases.World Chinese Journal of Digestology,2007(36):3856-3859.